CLINICAL TRIAL: NCT00638950
Title: Long-term Moderate Intervention With n-3 LC-PUFA-supplemented Dairy Products: Effects on Pathophysiological Biomarkers in Rheumatoid Arthritis
Brief Title: A Long-term Moderate Intervention With n-3 LC-PUFA-supplemented Dairy Products in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Prof. Dr. G. Jahreis, Universitiy of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSEP_H16-04
Record Dates: First submitted 2008-02-29; First posted 2008-03-19 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2008-02

CONDITIONS: Rheumatoid Arthritis
Keywords: n-3 LC-PUFA; Rheumatoid arthritis; disease activity; inflammation; oxidative stress; immune system
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- n-3 LC-PUFA (Active Comparator)
  Interventions: Dietary Supplement: n-3 LC-PUFA

INTERVENTIONS:
Dietary Supplement: n-3 LC-PUFA — Patients received about 40 g fat daily (200 g yoghurt with 3.8% fat, 30 g cheese with about 50% fat in the dry matter, and 20-30 g butter). The milk fat was partially exchanged by special oils. The daily dose of n-3 FA amounted to 2.4 g, consisting of 1.1 g ALA, 0.7 g EPA, 0.1 g DPA, and 0.4 g DHA.
  Arms: n-3 LC-PUFA
Dietary Supplement: Placebo — The placebo products were commercial dairy products with comparable fat contents.
  Arms: Placebo

SUMMARY:
The effects of n-3 LC-PUFA-supplemented dairy products on inflammation and immunological parameters, biomarkers of oxidative stress, serum lipids, and disease activity were determined in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Recent studies suggest that n-3 LC-PUFA may improve cardiovascular and inflammatory diseases.

As a precondition for participating in this study, the subjects were provided information in writing and verbally about the details of the study. Informed consent was obtained from all volunteers. Before the beginning of the study, all participants were subject to a medical examination in the Clinic for Rheumatology (Internal Medicine III, Friedrich Schiller University, Jena). The RA was diagnosed according to the 1987 revised criteria of the American Rheumatism Association (ARA). Severity of disease activity was evaluated by using the disease activity score DAS 28.

Forty five subjects (43 f, 2 m) were randomly divided into two groups to carry out a double-blind, placebo-controlled cross-over study.

The study consisted of two investigation periods of 12 weeks, with an eight-week washout period in between. Patients received about 40 g fat daily (200 g yoghurt with 3.8% fat, 30 g cheese with about 50% fat in the dry matter, and 20-30 g butter). The milk fat was partially exchanged by special oils with high amounts of eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA), and alpha linoleic acid (ALA). The daily dose of n-3 FA amounted to 2.4 g, consisting of 1.1 g ALA, 0.7 g EPA, 0.1 g DPA, and 0.4 g DHA. The placebo products were commercial dairy products with comparable fat contents.

Venous blood and 24h urine were collected at the beginning and at the end of each period. The DAS 28 score was assessed at the beginning and the end of each period, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Clear diagnosis of Rheumatoid Arthritis
* Patients receiving nonsteroidal anti-inflammatory drugs (NSAID) or corticosteroids (max. 15 mg/d) or both were eligible if dosage had been stable for at least 4 weeks before day 1 of the study and remained below this limit throughout the study
* Patients on disease-modifying antirheumatic drugs (DMARD) had to be on a constant dosage for at least 8 weeks before and throughout the study

Exclusion Criteria:

* Subjects with gastrointestinal or metabolic diseases, alcohol abuse, taking dietary supplements (e. g. fish oil capsules), known allergies or foodstuff indigestibility
* patient's request, serious infections, inadequate control of arthritis symptoms (over 50% increase of the number of swollen or tender joints), reinstitution of therapy with DMARD, or if patient compliance with the study protocol was doubtful.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-09; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
disease activity score DAS28 | 12 weeks
inflammatory markers (c-reactive protein, erythrocyte sedimentation rate) | 12 weeks

SECONDARY OUTCOMES:
cellular and humoral immunological parameters (CDs) | 12 weeks
COX expression | 12 weeks
biomarkers of oxidative stress (8-iso-prostaglandin F2α, 15-keto-dh prostaglandin F2α, 8-oxo-deoxy-guanosine) | 12 weeks
hydroxypyridinium crosslinks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — University of Jena, Dept. of Nutritional Physiology
Locations (1):
- University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Background] Dawczynski C, Schubert R, Hein G, Muller A, Eidner T, Vogelsang H, Basu S, Jahreis G. Long-term moderate intervention with n-3 long-chain PUFA-supplemented dairy products: effects on pathophysiological biomarkers in patients with rheumatoid arthritis. Br J Nutr. 2009 May;101(10):1517-26. doi: 10.1017/S0007114508076216. Epub 2009 Feb 27. PMID 19245735